CLINICAL TRIAL: NCT00410306
Title: International, Multi-center Post Authorization Surveillance Study on the Use of Nebido® to Assess Tolerability and Treatment Outcomes in Daily Clinical Practice (IPASS Nebido)
Brief Title: Use of Nebido® to Assess Tolerability and Treatment Outcomes in Daily Clinical Practice
Acronym: IPASS Nebido
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Medical Affairs Therapeutic Area Head, Bayer Schering Pharma AG
Other Study IDs: 14203; 2005/00888; MP-04199; NE0601; 39732
Record Dates: First submitted 2006-12-11; First posted 2006-12-12 (Estimated); Last update posted 2010-09-24 (Estimated); Status verified 2010-09

CONDITIONS: Male; Hypogonadism
Keywords: Hypogonadism; Nebido; Testosterone; Observational Study
MeSH Terms: conditions — Hypogonadism | interventions — testosterone undecanoate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Testosterone Undecanoate (Nebido, BAY86-5037)

INTERVENTIONS:
Drug: Testosterone Undecanoate (Nebido, BAY86-5037) — Patients from routine practice

SUMMARY:
This is an observational study with a drug called Nebido, a new testosterone replacement therapy, which is available for the treatment of male hypogonadism. The benefit and safety of Nebido have already been thoroughly evaluated through well controlled clinical trials. The main purpose of this observational study is to confirm the established safety profile of Nebido in daily clinical practice.

DETAILED DESCRIPTION:
The study has previously been posted by Schering AG, Germany. Schering AG, Germany has been renamed to Bayer Schering Pharma AG, Germany. Bayer Schering Pharma AG, Germany is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Male hypogonadal patients eligible for long-term testosterone therapy who have newly been prescribed Nebido® in accordance with the terms of the marketing authorization

Exclusion Criteria:

* Patients presenting with contraindications as stated in the product information

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from routine practice
Sampling Method: Non-Probability Sample
Enrollment: 1493 (Actual)
Dates: Start 2006-10; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Adverse events, adverse drug reactions, patient reported tolerability | during 4 injection intervals

SECONDARY OUTCOMES:
Change in laboratory values (total testosterone, estradiol, SHGB, FSH, LH) from baseline to end of observation | after 4 injection intervals
Change in subjective assessment of the patient (overall sexual desire/libido, vigor/vitality, mood, ability to concentrate) from baseline to end of observation | after 4 injection intervals
Change in intensity of symptoms or disorders associated with low testosterone (hot flushes or excessive sweating, sleep disturbances, decreased physical strength and erectile dysfunction) from baseline to end of observation | after 4 injection intervals
Patient reported outcome at end of observation (satisfaction with current androgen therapy, comparison to previous androgen therapy, if applicable) | after 4 injection intervals
Treatment continuation rate | after 4 injection intervals
Vital signs and anthropometric measurements (Blood pressure, heart rate, weight and waist circumference) | during 4 injection intervals
Laboratory values (PSA, hemoglobin, hematocrit, HbA1C, T-chol, HDL-chol, LDL-chol, triglycerides) | during 4 injection intervals
Digital rectal examination | during 4 injection intervals

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (33):
- Many Locations, Australia
- Many Locations, Austria
- Many Locations, Bulgaria
- Many Locations, Colombia
- Many Locations, Czechia
- Many Locations, Estonia
- Many Locations, Germany
- Many Locations, Hong Kong
- Many Locations, Indonesia
- Many Locations, Italy
- Many Locations, Jordan
- Many Locations, Kazakhstan
- Many Locations, Latvia
- Many Locations, Lebanon
- Many Locations, Lithuania
- Many Locations, Malaysia
- Many Locations, Malta
- Many Locations, Mexico
- Many Locations, Moldova
- Many Locations, North Macedonia
- Many Locations, Philippines
- Many Locations, Romania
- Many Locations, Russia
- Many Locations, Saudi Arabia
- Many Locations, Singapore
- Many Locations, Slovenia
- Many Locations, South Korea
- Many Locations, Spain
- Many Locations, Taiwan
- Many Locations, Thailand
- Many Locations, Turkey (Türkiye)
- Many Locations, Ukraine
- Many Locations, United Kingdom